CLINICAL TRIAL: NCT03709498
Title: Nutritional Status as a Prognostic Marker of Risk and Outcome in Patients Admitted to Hospital With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Nutritional Status in Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Dimitrios Karayiannis, Clinical Dietitian, Department of Clinical Nutrition and Metabolism, Evangelismos Hospital
Other Study IDs: 53/27-01-2016
Record Dates: First submitted 2018-10-09; First posted 2018-10-17 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Diet; Nutritional Status; Acute Exacerbation; Phase Angle
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross sectional observation study of body composition in COPD patients consecutively hospitalized with acute exacerbation.

DETAILED DESCRIPTION:
Skeletal muscle dysfunction and changes in body composition are important extra-pulmonary manifestations of chronic obstructive pulmonary disease (COPD) that occur in all stages of disease and are associated with poor outcome. In patients with COPD, bioelectrical impedance analysis (BIA) has usually been used to estimate fat-free mass (FFM) and body composition through predictive equations. Very few studies had focused on raw BIA data. The aim of this study is first describe the measurement of phase angle in patients with with acute exacerbation and second to determine the validity of phase angle in this group by assessing its relationship with established markers of function, disease severity and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of COPD based on history
* Hospitalization with acute COPD exacerbation

Exclusion Criteria:

* Patients with history of recent surgery (major) and trauma (major)
* Patients with concomitant disease that might alter nutritional status (heart disease, cirrhosis, uncontrolled diabetes, chronic renal failure, uncontrolled cor pulmonale).
* Contraindication to BIA including an implanted pacemaker, defibrillator or joint prosthesis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with COPD according to Global Initiative for Chronic Obstructive Lung Disease (GOLD)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Phase Angle | 1 month
  The evaluation of phase angle will be performed by means of the electric bioimpedance apparatus. The measurements will be obtained with the patient in dorsal decubitus, barefoot, with the lower limbs slightly apart and without metal objects attached to the body, with electrodes placed on the right hand and foot.

SECONDARY OUTCOMES:
Change in Forced vital capacity (FVC) | 1 month
  Secondary endpoint will be the correlation between FVC and muscle mass.
Correlation between phase angle and serum CRP levels. | 1 month
  Detect the serum CRP levels and then analyze the correlation between CRP and phase angle measurement.
Forced expiratory flow volume in one second (FEV1). | 1 month
  Forced expiratory flow volume in one second following standards recommended by European Respiratory Society and correlation with muscle mass.
Length of Hospital Stay (LOS) | 1 month
  Duration of Hospital Stay
Phase Angle | 2 months
  The evaluation of the phase angle will be performed by means of the electric bioimpedance apparatus. The measurements will be obtained with the patient in dorsal decubitus, barefoot, with the lower limbs slightly apart and without metal objects attached to the body, with electrodes placed on the right hand and foot.
Body Composition | 1 month.
  Body composition will be assessed using bioelectrical impedance analysis (In Body 720, Biospace) at a standardized time after breakfast. Bioelectrical impedance analysis (BIA) is a simple, safe, non-invasive method to measure assess lean (e.g., muscle) vs. fat body compartments. Fat-free mass will be calculated by using disease-specific equations as described by Schols. Fat mass will then be calculated as total body weight minus fat-free mass. Such BIA measurements are accurate, comparable to other techniques used to assess body composition, and have been validated in patients with acute excerbation of COPD

CONTACTS AND LOCATIONS:
Overall Officials: Sotirios Kakkavas, MD, PhD, Principal Investigator — Pulmonary Medicine Dept, Evangelismos Hospital,
Locations (1):
- Department of Nutrition and Dietetics, Evaggelismos Hospital, Athens, Kolonaki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] S. Kakavas, D. Karayiannis, A. Papanikolaou, A. Baschali, M. Sarantidou, A. Karachaliou, A. Karli, Z. Mastora, M. Palavra, G. Boulbasakos. Bioelectrical Impedance Analysis Phase Angle as a Prognostic Marker for Outcome in Patients Admitted in Hospital with Acute Exacerbation of Chronic Obstructive Pulmonary Disease. Clinical Nutrition 36:S101, 2017